CLINICAL TRIAL: NCT02076724
Title: Reinforcement of the Abdominal Wall With Acellular Dermal Matrix (Strattice™) After Breast Reconstruction With the Pedicled TRAM-flap
Brief Title: Reinforcement of the Abdominal Wall After Breast Reconstruction With the Pedicled TRAM-flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: LifeCell (Industry); Novo Nordisk A/S (Industry); University of Aarhus (Other)
Responsible Party: Principal Investigator, Mette Eline Brunbjerg, MD, MD, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VEK 1-10-72-10-13
Record Dates: First submitted 2014-02-26; First posted 2014-03-04 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Abdominal Donor-site
Keywords: Abdominal donor-site; Breast reconstruction; Synthetic mesh; Biological mesh

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biological mesh (Strattice Firm) (Experimental): Strattice Firm is inserted using inlay technique as reinforcement of the abdominal wall where the anterior rectus fascia has been excised.
  Interventions: Device: Biological mesh
- Synthetic mesh (Prolene) (Experimental): Prolene mesh is inserted using inlay technique as reinforcement of the abdominal wall where the anterior rectus fascia has been excised.
  Interventions: Device: Synthetic mesh

INTERVENTIONS:
Device: Biological mesh
  Other Names: Strattice Reconstructive Tissue Matrix Firm, LifeCell Corp.
  Arms: Biological mesh (Strattice Firm)
Device: Synthetic mesh
  Other Names: Prolene mesh, Ethicon
  Arms: Synthetic mesh (Prolene)

SUMMARY:
The purpose of this study is to compare two methods for reinforcement of the abdominal donor-site after breast reconstruction with the pedicled TRAM-flap. Reinforcement of the abdominal donor-site is performed, after randomization, with either a porcine derived biological mesh or a synthetic mesh. The patient and the investigator is blinded.

The aim is to identify the most optimal method for reinforcement of the abdominal donor-site and thereby contribute to fast and complete rehabilitation of women undergoing breast reconstruction with the pedicled TRAM-flap after surgical removal of the breast tissue due to breast cancer, precursors to breast cancer or an increased risk of developing breast cancer and thereby following preventive removal of the breast tissue.

The patients visit the outpatient clinic 4, 12 and 24 months after operation and abdominal wall function, the donor site morbidity, the frequency of postoperative complications, the aesthetic appearance of the reconstructed breast and the abdominal wall and costs are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Immediate or delayed breast reconstruction using the pedicled TRAM-flap
* Older than 18 years of age
* Understand enough Danish to comprehend the given information and to complete the study questionnaire
* Verbal and written informed consent

Exclusion Criteria:

* Current smokers
* Not eligible patients, assessed by surgeon
* High level of co-morbidity, assessed by surgeon or anesthesiologist

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Abdominal wall function change | Change from before surgery to 12 and 24 months after surgery
  Strength of abdominal wall is assessed by a standardized physical examination developed in collaboration with physiotherapists. A dynamometer is used to get an exact value of muscle strength.

SECONDARY OUTCOMES:
Abdominal donor site morbidity | 24 months
  Bulge
  * Definition: visible abdominal contour abnormality, without the presence of a fascial defect, with or without the need for surgical correction.
  * Assessed after 3-4, 12 and 24 months by clinical examination and after 12 and 24 months by CT scanning including the Valsalva maneuver
  Hernia
  * Definition: abdominal wall bulge with the presence of a palpable fascial defect and/or a fascial defect found during an additional correcting surgical procedure or by CT scanning.
  * Assessed after 3-4, 12 and 24 months by clinical examination and after 12 and 24 months by CT scanning including the Valsalva maneuver
  Abdominal donor site correction procedure (within 24 months)
  Pain/ discomfort
  * Assessed after 3-4, 12 and 24 months by
  * DoloTest®
  * Study specific questionnaire regarding postoperative assessment of abdominal pain/ discomfort including effect on daily life activities and ability to perform sport
Aesthetics at the abdominal wall | 24 months
  Study specific questionnaire regarding postoperative assessment of the outcome including:
  * Overall satisfaction with the appearance of the abdominal donor site
  * Satisfaction regarding placement and the appearance of the umbilicus
  Investigators assessment of the abdominal donor site including:
  * Visual bulging of the lower abdomen
  * Placement and appearance of the umbilicus
  * Appearance of the scar
Costs | 24 months
  National health insurance rate Cost of Strattice (LifeCell), Prolene mesh (Ethicon) Operation time Hospitalization Time to return to work / Duration of sick leave Post-reconstruction procedures to address complications at the abdominal donor site.
Postoperative complications | Acute <1 month, ≥ 1 month-24 months
  Hematoma requiring surgical intervention. Cellulitis/ wound infection not requiring surgical intervention but treatment with antibiotics.
  Infection requiring surgical intervention. Seroma requiring intervention Donor site necrosis (present necrosis - excluding epidermolysis, in the umbilical area or in the remaining abdominal skin and subcutaneous tissue requiring surgical intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Mette Eline Brunbjerg, MD, Principal Investigator — Aarhus University Hospital and Aarhus University
Locations (1):
- Department of Plastic and Reconstructive Surgery, Aarhus University Hospital, Aarhus C, Aarhus, Denmark